CLINICAL TRIAL: NCT04137692
Title: Red Blood Cell Exchange Transfusion as a Novel Treatment for GLUT1 Deficiency Syndrome
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: PI is transferring institutions.
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 24-07027753; RM1NS133593 (NIH)
Record Dates: First submitted 2019-10-08; First posted 2019-10-24 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Glucose Transporter Type 1 Deficiency Syndrome; GLUT1DS1
Keywords: G1D; Glucose transporter
MeSH Terms: conditions — Glut1 Deficiency Syndrome | interventions — Erythrocyte Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Red Blood Cell Transfusion (Experimental): Patients will undergo isovolemic hemodilution-red cell exchange (IHD- RBCx) with up to 10 units of red cell antigens (Rh group, Kell, Duffy, Kidd blood group antigens) matched normal donor red cells to replace a target of 70% of the patient's red cells with donor red cells.
  Interventions: Other: Red Blood Cell Transfusion

INTERVENTIONS:
Other: Red Blood Cell Transfusion — The procedure will be performed as an outpatient according to protocols established for sickle cell anemia patients. Two IVs are placed for the purposes of transfusion, one for draw and one for return. Patients will undergo isovolemic hemodilution-red cell exchange (IHD- RBCx) with up to 10 units of red cell antigens (Rh group, Kell, Duffy, Kidd blood group antigens) matched normal donor red cells to replace a target of 70% of the patient's red cells with donor red cells.Total time of procedure: approximately 150 minutes.

SUMMARY:
Pathogenic mutations of the brain glucose transporter type I lead to glucose transporter deficiency syndrome (G1D), which is most often associated with medication-refractory epilepsy and movement dysfunction. At present, G1D is only alleviated by interventions such as the ketogenic diet, which can be poorly tolerated and afford only an incomplete restoration of neural function. A better understanding of G1D can uncover new fundamental aspects of brain function while facilitating the development of new therapies aimed to restore brain metabolism and excitability. We will conduct a mechanistic trial that will utilize a mechanism-testing framework broadly applicable to metabolic interventions. The trial will investigate red blood cell exchange (i.e., the replacement of human G1D circulating red cells, which are deficient in GLUT1) with healthy donor cells as a novel means to augment blood-to-brain glucose transport. The hypothesis is that electroencephalography post treatment will display an increase in beta brain activity. Additional measures of brain activity will also be secondarily tested.

DETAILED DESCRIPTION:
Glucose Transporter 1 (GLUT1) is a protein that helps move glucose (sugar) into cells. Most tissues in the body have only small amounts of this protein. Red blood cells, however, have very large amounts of GLUT1, far more than they need for their own energy use. Because of this, red blood cells can take in and carry glucose at extremely high rates, much higher than they can actually use themselves. Some scientists believe that red blood cells may serve as a temporary storage system for glucose, especially when blood sugar levels are low. If this idea can be proven, it would change how we understand an important part of human biology.

This study may also lead to new treatment options for people with Glucose Transporter Type 1 Deficiency (G1D). G1D is a condition where the brain does not get enough glucose because the GLUT1 protein does not work properly. Right now, the only treatment is the ketogenic diet. This diet helps some patients with seizures, but it does not work well for long-term brain development or overall health, so better treatments are needed. It is usually believed that G1D mainly affects the cells in the brain's blood vessels, which help control what gets into the brain. However, many G1D patients also have low levels of GLUT1 in their red blood cells, meaning their red blood cells may not carry enough glucose. This may also play a role in the disease. Animal models, like mice with GLUT1 deficiency, do not accurately mimic the human condition, so they cannot fully answer this question. Red blood cell exchange (RBCx) is already used safely and at reasonable cost for patients with sickle cell disease to prevent strokes and blood vessel problems. Because RBCx replaces a person's red blood cells with donor cells, it could be a promising new approach for treating G1D.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female
2. Age 16 years to 80 years old.
3. Diagnosed with genetically confirmed glucose transporter type 1 disorder
4. Patients not currently receiving ketogenic dietary therapy, due to failure of this diet to achieve seizure remission or due to patient preference, including compliance or tolerance issues.
5. Subjects must be able to provide informed consent for themselves or have a parent or legally authorized representative (LAR) provide permission if the subject is a minor or lacks capacity to consent.
6. Spanish and English speakers will be eligible for participation. Spanish-speaking participants may be enrolled, and the study team is equipped to conduct the consent process in Spanish. The Principal Investigator (PI) is fluent in Spanish and will conduct the consent process in Spanish when applicable.
7. IHD-RBCx is determined to be a safe and appropriate procedure for the subject by the transfusion medicine physician based on clinical and laboratory assessment.

Exclusion Criteria:

1. Currently on the ketogenic diet or taking triheptanoin (C7) oil
2. No genetic confirmation of G1D diagnosis
3. Unable to return for follow up visits
4. Weak peripheral veins, such that IV placement is contraindicated (required for transfusion)
5. Serious chronic medical conditions, such as congestive heart failure, renal failure, liver failure, or any other medical conditions that preclude large volume transfusions.
6. Patients currently pregnant or breast-feeding are excluded from participating in this research. Patients who plan on getting pregnant during this research or who are unwilling to use birth control, including abstinence, during the course of this research are also excluded due to safety concerns for the fetus.
7. An evaluation by the transfusion physician as to whether IHD-RBCx is a safe option will be part of the screening assessment. If IHD-RBCx is deemed unsafe based on laboratory parameters such as a low red blood cell count, then the subject will not be eligible to participate in this study.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2027-09 (Estimated); Primary Completion 2030-08 (Estimated); Study Completion 2031-08 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in electroencephalography (EEG) measures during transfusion. | Baseline: During Transfusion
  Electroencephalography measures number of seizures recorded during the transfusion. Number of seizures will be assessed using standard observation of the electroencephalogram (EEG).
Change from baseline in electroencephalography (EEG) measures 60 days after transfusion. | Baseline - 60 Days After Transfusion
  Electroencephalography measures number of seizures recorded 60 days after the transfusion. Number of seizures will be assessed using standard observation of the electroencephalogram (EEG).

SECONDARY OUTCOMES:
Change from baseline in Peabody Picture Vocabulary Test (PPVT) standard scores immediately after transfusion | Baseline - Immediately after transfusion
  The Peabody Picture Vocabulary Test (PPVT) measures receptive vocabulary skills. Total scores range from 20 to 160, with higher scores indicating stronger receptive language ability.
Change from baseline in Peabody Picture Vocabulary Test (PPVT) standard scores 60 days after transfusion | Baseline - 60 days after transfusion
  The Peabody Picture Vocabulary Test (PPVT) measures receptive vocabulary skills. Total scores range from 20 to 160, with higher scores indicating stronger receptive language ability.
Change from baseline in Expressive Vocabulary Test (EVT) standard scores immediately after transfusion | Baseline - Immediately after transfusion
  The Expressive Vocabulary Test (EVT) evaluates expressive vocabulary and word retrieval abilities. Total Standard scores typically range from 20 to 160, with higher scores indicating stronger expressive language skills.
Change from baseline in Expressive Vocabulary Test (EVT) standard scores 60 days after transfusion | Baseline - 60 days after transfusion
  The Expressive Vocabulary Test (EVT) evaluates expressive vocabulary and word retrieval abilities. Total Standard scores typically range from 20 to 160, with higher scores indicating stronger expressive language skills.
Change from Baseline in T-scores on the Connors Continuous Performance Test Immediately After Transfusion | Baseline - Immediately after transfusion
  T-scores will be obtained from the Connors Continuous Performance Test (CPT). Minimum T-score is <30 and maximum is 90. For the Hit Reaction Time domain, higher T-scores indicate slower reaction time. For detectability, omissions, commissions, and perseverations, higher T-scores indicate elevated performance.
Change from Baseline in T-scores on the Connors Continuous Performance Test 60 Days After Transfusion | Baseline - 60 days after transfusion
  T-scores will be obtained from the Connors Continuous Performance Test (CPT). Minimum T-score is <30 and maximum is 90. For the Hit Reaction Time domain, higher T-scores indicate slower reaction time. For detectability, omissions, commissions, and perseverations, higher T-scores indicate elevated performance.
Number of participants immediately after transfusion with erythrocyte Glut1 levels increased by over 40% from baseline | Immediately after transfusion
  Baseline erythrocyte Glut1 levels are used as the reference point. This measure captures the number of participants whose Glut1 levels increase by more than 40% immediately after transfusion compared to their baseline value.
Number of participants 60 days after transfusion with erythrocyte Glut1 levels increased by over 40% from baseline | 60 days after transfusion
  Baseline erythrocyte Glut1 levels are used as the reference point. This measure captures the number of participants whose Glut1 levels increase by more than 40% 60 days after transfusion compared to their baseline value.
Change from Baseline in General Medical & Neurological Examination 60 Days After Transfusion | Baseline - 60 days after transfusion
  This measure assesses change from baseline in the standardized clinical physical examination, which includes 12 domains scored as normal or abnormal. Minimum total score is 0. Maximum total score is 76. Higher total scores indicate a more normal examination and better outcomes, while lower scores indicate more abnormalities.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Pascual, MD, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose.

REFERENCES:
- [Background] Lee EE, Ma J, Sacharidou A, Mi W, Salato VK, Nguyen N, Jiang Y, Pascual JM, North PE, Shaul PW, Mettlen M, Wang RC. A Protein Kinase C Phosphorylation Motif in GLUT1 Affects Glucose Transport and is Mutated in GLUT1 Deficiency Syndrome. Mol Cell. 2015 Jun 4;58(5):845-53. doi: 10.1016/j.molcel.2015.04.015. Epub 2015 May 14. PMID 25982116
- [Derived] Wang RC, Lee EE, De Simone N, Kathote G, Primeaux S, Avila A, Yu DM, Johnson M, Good LB, Jakkamsetti V, Sarode R, Holland AA, Pascual JM. Red blood cells as glucose carriers to the human brain: Modulation of cerebral activity by erythrocyte exchange transfusion in Glut1 deficiency (G1D). J Cereb Blood Flow Metab. 2023 Mar;43(3):357-368. doi: 10.1177/0271678X221146121. Epub 2022 Dec 15. PMID 36523131